CLINICAL TRIAL: NCT03566108
Title: A Prospective, Randomized Clinical Trial to Compare Vestibular Incision Supraperiosteal Tunnel Access (VISTA) and Sulcular Tunnel Access Procedures With Coronally Advanced Flap (CAF) and Acellular Dermal Matrix (ADM).
Brief Title: To Compare Two Commonly Used Soft Tissue Grafting Techniques to Achieve Coronal Flap Advancement and Root Coverage
Acronym: VISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maria L. Geisinger, DDS, MS, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300001591; UAB Periodontology (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2018-05-14; First posted 2018-06-21 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Gingival Recession
Keywords: Gingival phenotype; Keratinized gingiva; Gingival recession; Soft tissue recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VISTA (Experimental): VISTA incision with CAF and ADM
  Interventions: Procedure: VISTA
- Sulcular Tunnell access (Active Comparator): Sulcular tunnel surgery with CAF and ADM
  Interventions: Procedure: STA

INTERVENTIONS:
Procedure: VISTA — Vestibular incision supraperiosteal tunnel access (VISTA) incision will be performed on all individuals in this arm of the study to facilitate coronal advancement of the gingival flap and placement of acellular dermal matrix
  Arms: VISTA
Procedure: STA — Sulcular tunnel access incision will be performed on all individuals in this arm of the study to facilitate coronal advancement of the gingival flap and placement of acellular dermal matrix
  Arms: Sulcular Tunnell access

SUMMARY:
This study will compare two incision designs to allow for coronal gingival/mucosal flap advancement and tissue augmentation with acellular dermal matrix (ADM) graft around teeth with gingival recession and a lack of adequate keratinized gingiva.

To the investigators knowledge, these two techniques have not been compared for differences in clinical (amount of root coverage, tissue thickness, and esthetics) and patient-centered outcomes (pain, swelling, change in daily activities) in a controlled study.

DETAILED DESCRIPTION:
Research data and daily clinical observations reveal that teeth with gingival recession and a lack of adequate keratinized tissue (KT) are more prone to persistent gingival inflammation, dentinal sensitivity, radicular (root) caries (tooth decay), faster periodontal attachment loss, and compromised plaque control. Soft tissue grating (by various techniques) aims at changing the quality, quantity and placement of the soft tissue around teeth by covering exposed root surfaces and creating or increasing the zone of keratinized mucosa (KM) surrounding the affected teeth. Both techniques tested have shown good clinical outcomes with regard to root coverage, but clinical reports of the VISTA technique and other similar techniques suggest that patients experience a decrease in site morbidity and discomfort post-operatively. This study will compare two surgical incision designs used in conjunction with coronally advanced flap (CAF) and acellular dermal matrix (ADM)

Specific aims for this project include the evaluation of:

* Percentage of root coverage at 6 and 12 months following grafting with VISTA and sulcular tunnel access with ADM
* KT width at 6 and 12 month following grafting with VISTA and sulcular tunnel access with ADM
* Change in tissue thickness of the grafted sites at 6 and 12 months
* Practitioner-assessed esthetic outcomes using a standardized pink esthetic scale (PES) at 6 and 12 months postoperatively
* Patient-assessed esthetic outcomes at 6 and 12 months post-operatively
* Patient centered outcomes including pain, bleeding, swelling, change in daily activities at 1 week and 1 month postoperatively

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* At least 18 years old
* Must be a patient of the UAB Dental School
* Able to read and understand informed consent document
* One or more adjacent teeth (up to four) with Miller class I or II gingival recession defects and less than or equal to 2mm of KT at each site to be treated.
* Presence of periodontally healthy, non-carious neighboring teeth, healthy implants or edentulous ridges on either side of the involved site(s)
* No anticipated need for restorative care at the teeth to be treated during the study period.

Exclusion Criteria:

* Non-English speaking
* Less than 18 years old
* Smokers/tobacco users (>10 cigarettes/day)
* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing
* Presence of active periodontal disease or radiographic interproximal bone loss or tooth malposition, which would yield a Miller class III or IV categorization for the recession defect.
* Presence of frenulae or other soft tissue anomalies at the site(s) to be treated that, in the opinion of the investigators, will interfere with successful access and treatment of the soft tissue defects.
* Previous soft tissue grafting at the site(s) to be treated

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Geisinger, DDS, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be shared with other researchers outside of our research laboratory group.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 9 participants enrolled in the study, 2 (VISTA), 1 (STA) and 6 (VISTA and STA). Randomization was performed by site in the mouth (teeth) to receive either VISTA intervention or STA intervention. As a result, some participants received one of the 2 interventions either VISTA or STA if they only had one qualifying site (teeth), while other participants received both interventions if they had multiple sites that are met the inclusion criteria. Total VISTA sites=13, total STA sites=16.
Units Other Than Participants: site (teeth)
Groups:
- VISTA Only: VISTA incision with CAF and ADM
- Sulcular Tunnel Access (STA) Only: Sulcular tunnel surgery with CAF and ADM
- VISTA + STA: STA; VISTA + STA; VISTA: Both VISTA and STA (at different sites in the same patient)
Period: Overall Study
Arm/Group | VISTA Only | Sulcular Tunnel Access (STA) Only | VISTA + STA: STA | VISTA + STA; VISTA
Started | 2; 3 site (teeth) | 1; 1 site (teeth) | 6; 15 site (teeth) | 6; 10 site (teeth)
Completed | 2; 3 site (teeth) | 1; 1 site (teeth) | 6; 15 site (teeth) | 6; 10 site (teeth)
Not Completed | 0; 0 site (teeth) | 0; 0 site (teeth) | 0; 0 site (teeth) | 0; 0 site (teeth)

BASELINE CHARACTERISTICS:
Units Other Than Participants: site (teeth)
Groups:
- Sulcular Tunnel Access (STA): Sulcular tunnel surgery with CAF and ADM
- VISTA + STA: Both VISTA and STA (at different sites in the same patient)
- Total: Total of all reporting groups
Arm/Group | VISTA | Sulcular Tunnel Access (STA) | VISTA + STA | Total
Number analyzed (Participants) | 2 | 1 | 6 | 9
Number analyzed (site (teeth)) | 3 | 1 | 25 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 5 | 8
  >=65 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3
  Male | 1 | 1 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 1 | 6 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: KT Width at 6 Month Following Grafting With VISTA and Sulcular Tunnel Access With ADM
Description: Compare the increase in keratinized tissue (KT) between two incision designs for root coverage and tissue augmentation.
Time Frame: From baseline to 6 months
Population: VISTA group has 2 participants who only received VISTA (number of sites=3) and has 6 participants who received VISTA (number of sites=10) total VISTA sites =13. STA group has 1 participant who only received STA (number of site=1) and has 6 participants who received VISTA and STA (number of sites=15) total STA sites=16).
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: site (teeth)
Arm/Group | VISTA | Sulcular Tunnell Access
Number analyzed (Participants) | 8 | 7
Number analyzed (site (teeth)) | 13 | 16
mm | 3.15 (0.27) | 2.23 (0.25)

2. Secondary Outcome: Change in Tissue Thickness at Gingival Margin of the Grafted Sites at 6 Months With ADM
Description: Using a periodontal probe, soft tissue thickness will be measured (in mm) and compared between VISTA and STA following soft tissue grafting.
Time Frame: From baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: site (teeth)
Arm/Group | VISTA | Sulcular Tunnell Access
Number analyzed (Participants) | 8 | 7
Number analyzed (site (teeth)) | 13 | 16
mm | 1.04 (0.045) | 0.95 (0.031)

3. Secondary Outcome: Change in Tissue Thickness 5mm Apical to Gingival Margin of the Grafted Sites at 6 Months With ADM
Description: as for outcome 2
Time Frame: From baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: site (teeth)
Arm/Group | VISTA | Sulcular Tunnell Access
Number analyzed (Participants) | 8 | 7
Number analyzed (site (teeth)) | 13 | 16
mm | 1.38 (0.14) | 1.12 (0.1)

4. Secondary Outcome: Assessed Esthetic Outcomes Using a Standardized Pink Esthetic Scale (PES) at 6 Months Postoperatively
Description: Assess esthetic outcomes using an established Periodontal Esthetic Score (PES). This score evaluates the color of the gum utilizing 5 subscales ranging from 0 (worse) to 2 (better) allowing for a summed total score of 10.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: site (teeth)
Arm/Group | VISTA | Sulcular Tunnell Access
Number analyzed (Participants) | 8 | 7
Number analyzed (site (teeth)) | 13 | 16
score on a scale | 7.41 (0.28) | 7.31 (0.29)

ADVERSE EVENTS:
Time Frame: baseline to 6 months
Groups:
- VISTA Only: VISTA incision with CAF and ADM
  VISTA: Vestibular incision supraperiosteal tunnel access (VISTA) incision will be performed on all individuals in this arm of the study to facilitate coronal advancement of the gingival flap and placement of acellular dermal matrix
- Sulcular Tunnell Access(STA) Only: Sulcular tunnel surgery with CAF and ADM
  STA: Sulcular tunnel access incision will be performed on all individuals in this arm of the study to facilitate coronal advancement of the gingival flap and placement of acellular dermal matrix
- VISTA+STA: Both VISTA and STA (at different sites in the same patient)
Arm/Group | VISTA Only | Sulcular Tunnell Access(STA) Only | VISTA+STA
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/6
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/6

LIMITATIONS AND CAVEATS:
Randomization was performed by site (teeth) due to challenges recruiting sufficient participants for both arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT03566108/Prot_SAP_000.pdf